## **Informed Consent Form**

Title: Short-Term Effects of Acupuncture on Balance and Quality of Life in Women with Migraine: A Pilot Study

ClinicalTrials.gov Identifier (NCT Number):

Responsible Party: Klaipėda University, Holistic Medicine and Rehabilitation Department

Principal Investigator: PhD Laura Zaliene, Klaipėda University

Document Date: 2025-08-25

Contact Information: +37067499009, laura.zaliene@ku.lt

- 1. **Purpose of the Study.** You are invited to take part in a research study. The purpose of this pilot study is to evaluate the short-term effects of acupuncture on balance and quality of life in women with migraine.
- 2. **Procedures** If you agree to participate, you will undergo a series of acupuncture sessions over a deRined period. Before and after the intervention, we will assess your balance, migraine intensity, and quality of life using validated questionnaires and stabilometric testing. Each session will last approximately [20 minutes].
- 3. **Possible Risks and Discomforts** Acupuncture is generally considered safe. Possible minor side effects include: Mild pain, redness, or bruising at the needle site Temporary dizziness or fatigue Rare allergic reactions to sterile needles
- 4. **Possible Benefits** You may experience reduced migraine symptoms, improved balance, and enhanced quality of life. However, these beneRits cannot be guaranteed.
- 5. **Voluntary Participation** Your participation is entirely voluntary. You may refuse to participate or withdraw from the study at any time, without giving a reason and without any consequences.
- 6. **Confidentiality** All data collected will be kept conRidential. Your identity will not be revealed in publications or presentations. Only anonymized data will be analyzed.
- 7. **Alternatives** Participation in this study is optional. You may choose not to participate and continue with your usual care.
- 8. **Compensation and Costs** There is no Rinancial cost to you. You will not receive payment for participation.
- 9. **Ethical Approval** This study has been approved by the Klaipė da University Bioethics Committee and follows the principles of the Declaration of Helsinki.
- 10. **Contact Informa4on** If you have questions about the study, please contact: Principal Investigator: [Name, contact details] If you have concerns about your rights as a participant, you may contact the Klaipė da University Bioethics Committee.

| 11. | 11. Consent Statement I have read and understood t | the information provided above. I have |
|---|---|---|
| | had the opportunity to ask questions, and they were an | nswered to my satisfaction. I voluntarily |
| | agree to participate in this study. | |

| 12. Participant's Name: | Signature: |
|-------------------------|------------|
| Date: | _ |
| 13.Investigator's Name: | Signature: |
| Date: | _ |